CLINICAL TRIAL: NCT04510883
Title: Usage and Health Effects of Embodied Conversational Agents Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); WAAG (Unknown); Roessingh Research and Development (Other); National Foundation for the Elderly (Unknown)
Responsible Party: Principal Investigator, Lean Kramer, Researcher, Wageningen University and Research
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 40-44300-98-110
Record Dates: First submitted 2020-07-13; First posted 2020-08-12 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Eating Behavior; Loneliness; Technology Use
Keywords: eHealth; Embodied Conversational Agent; Technology use
MeSH Terms: conditions — Feeding Behavior | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: An unblinded randomized controlled trial. Participants in the first cohort directly receive the intervention for 8 weeks. Participants in the second cohort receive the intervention after a waiting list condition of 4 weeks, serving as a control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACO (Experimental): Participants are asked to use the intervention for eight weeks.
  Interventions: Behavioral: PACO
- Waiting list + PACO (Other): Participants receive the same intervention, but only after a waiting period of four weeks.
  Interventions: Behavioral: Waiting list + PACO

INTERVENTIONS:
Behavioral: PACO — The intervention is a fully-automated web-based eHealth application in which two embodied conversational agents engage in dialogue with older adults in order to motivate them towards dietary behavior change and decrease loneliness. The application consists of five different modules, each one applying different behavior change techniques.
  Arms: PACO
Behavioral: Waiting list + PACO — Waiting list + PACO
  Arms: Waiting list + PACO

SUMMARY:
Rationale: Embodied Conversational Agents (ECAs), could be a highly effective medium to address health behaviour change among older adults. As compliance to health advice is important for positive health outcomes, successful design of persuasive ECAs can have huge health benefits. However, insights in the mechanisms underlying usage and health behaviour change via ECAs are lacking.

Objective: The objective is to unravel the mechanisms behind the use of an ECA intervention, and understand the mechanism behind the observed behaviour change

Study design: A randomized staggered-entry waitlist-controlled trial will be carried out.

Study population: The study population consist of Dutch-speaking older adults, who live independently, are without partner, are retired, 65+ and possess basic computer skills.

Intervention: The application PACO has been created for (and with) older adults with the goal to motivate them to improve their eating behaviour and decrease their feelings of loneliness.

Main study parameters/endpoints: The main study parameters are use, loneliness, and eating behaviour.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects are not exposed to any risks, nor have they any costs. They do have to fill in questionnaires and use the application. The duration and data collection moments are needed to gain a fine-grained understanding of the use, relationship development and health change process. For subjects, the main benefit is to gain insight in their health behaviour via the PACO-application. Although this might be experienced as confronting by some. The technology was developed based on sound theories, with input from the target group, so the investigators expect positive experiences and an improvement in participants loneliness and eating behaviour. However, this can only be proven after the study.

ELIGIBILITY:
Inclusion Criteria:

* Living independently at home
* Living without a partner
* No paid profession and at least 65 years of age
* Dutch speaking
* Able to use a tablet or computer
* Internet connection at home

Exclusion Criteria:

* Not willing to provide inform consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Logdata on use application | 8 weeks
  Amount of time spend on the application during the 8 weeks intervention period
Change in De Jong Gierveld Loneliness Scale | Four weeks before intervention to eight weeks
  Score from 1-5, higher score means a better outcome.
Change in eating behaviour based on 24 hours recall | Four weeks before intervention to eight weeks

SECONDARY OUTCOMES:
Enjoyment via affect scale | Eight weeks after intervention
  Pleasure in using the application. Score from 1-5, higher score means a better outcome.
Classic aesthetics Scale | Eight weeks after intervention
  The design of the application. Score from 1-7, higher score means a better outcome.
Concern for privacy scale | Four and eight weeks after intervention
  Concerns about sharing personal data, e.g.name and date of birth. Score from 1-7, higher score means a better outcome.
Active control scale | Eight weeks after intervention
  Control over the system, as perceived by the user. Score from 1-7, higher score means a better outcome.
System Usability Scale | Eight weeks after intervention
  Whether PACO is easy to use. Score from 1-5, higher score means a better outcome.
Perceived usefulness scale | Eight weeks after intervention
  Score from 1-5, higher score means a better outcome.
Rapport scale | Four weeks before intervention to eight weeks
  Relationship with the embodied conversational agent. Score from 1-5, higher score means a better outcome.
Brief Older People's Quality of Life Scake | Four weeks before intervention to eight weeks
  Score from 1-5, higher score means a better outcome.
Change in Basic Psychological Need Satisfaction and Frustration Scales | Four weeks before intervention to eight weeks
  Score from 1-5, higher score means a better outcome.

OTHER OUTCOMES:
Willingness to pay single questions | Eight weeks after intervention
  Willing to pay for PACO (y/n)
User experience via self-formulated open question | Four and eight weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emely de Vet, PhD, Principal Investigator — Wageningen University & Research
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the Data Management Plan, part of the data will be anonymized and made available in DANS-EASY with restricted access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available within 12 months after the end of the study.

REFERENCES:
- [Derived] Kramer LL, van Velsen L, Clark JL, Mulder BC, de Vet E. Use and Effect of Embodied Conversational Agents for Improving Eating Behavior and Decreasing Loneliness Among Community-Dwelling Older Adults: Randomized Controlled Trial. JMIR Form Res. 2022 Apr 11;6(4):e33974. doi: 10.2196/33974. PMID 35404255
- [Derived] Kramer LL, Mulder BC, van Velsen L, de Vet E. Use and Effect of Web-Based Embodied Conversational Agents for Improving Eating Behavior and Decreasing Loneliness Among Community-Dwelling Older Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jan 6;10(1):e22186. doi: 10.2196/22186. PMID 33404513